CLINICAL TRIAL: NCT00191945
Title: A Randomized Double-Blind, Placebo-Controlled Clinical Trial of Efficacy and Safety of Atomoxetine up to 12 Weeks in Newly Diagnosed Children and Adolescents Outpatients With Attention-Deficit/Hyperactivity Disorder
Brief Title: Efficacy and Safety of Atomoxetine in Children With Recent Diagnosis of Attention-Deficit/Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 8836; B4Z-XM-LYDM (Other: Eli Lilly and Company)
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2010-01-26 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2010-01

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atomoxetine (Experimental): atomoxetine: 0.5 mg/kg/day every day (QD),by mouth (PO) for 2 weeks, 1.2 - 1.4 mg/kg/day QD, PO for 10 weeks, then 1.2 - 1.4 mg/kg/day QD, PO for up to 1 year
  Interventions: Drug: Atomoxetine Hydrochloride
- Placebo (Placebo Comparator): placebo every day (QD), by mouth (PO) for 12 weeks,then possibility to switch to atomoxetine at 0.5 mg/kg/day QD, PO for 1 week, then to 1.2 - 1.4 mg/kg/day QD, PO for up to 1 year (open-label extension)
  Interventions: Drug: Atomoxetine Hydrochloride; Drug: placebo

INTERVENTIONS:
Drug: Atomoxetine Hydrochloride
  Other Names: LY139603; Strattera
Drug: placebo
  Arms: Placebo

SUMMARY:
Double blinded clinical trial placebo controlled in 153 children (planned enrollment) with recent diagnosis of ADHD. Patients will be randomized to atomoxetine or placebo arm (2:1). The double blinded period will last 12 weeks and the treatment open phase will last up to 1 year, and atomoxetine treatment will be administered.

A gatekeeper strategy will be employed for sequentially testing the secondary objectives.

ELIGIBILITY:
Inclusion Criteria:

1. Child or adolescent patients must be at least 6 years of age, but must not yet have reached their 16th birthday prior to Visit 1, when informed consent is obtained.
2. Patients must meet the Diagnostic and Statistical Manual for Mental Disorders, Fourth Edition Text Revision (DSM-IV-TR) diagnostic criteria for ADHD. For the purposes of this study the diagnosis of ADHD will be confirmed during Visit 1 by administering the K-SADS-PL. Patients must also have an ADHDRS-IV-Parent:Inv score at least 1.5 standard deviations above the age norm for their diagnostic subtype at both Visit 1 and Visit 2. In addition, they must have a CGI-ADHD-S score 4 at both Visit 1 and Visit 2.
3. Patients must have a newly diagnosed case of ADHD. Newly diagnosed case of ADHD means that a specialist (including pediatrician, child psychiatrist, or child neurologist) or child psychologist has diagnosed ADHD (according DSM-IV-TR or International Statistical Classification of Diseases and Related Health Problems [World Health Organisation; 10th Revision] [ICD 10] criteria) within 3 months prior to Visit 1.

Exclusion Criteria:

1. Patients with history of ADHD diagnosis longer than 3 months prior to Visit 1. Diagnosis of ADHD means that a specialist (including pediatrician, child psychiatrist, or child neurologist) or child psychologist has diagnosed ADHD (according DSM-IV-TR or ICD 10 criteria) and has registered it in medical records or verbally informed parents about this diagnosis.
2. Patients who weigh less than 20 kg at study entry (Visit 1). If a patient's weight changes after Visit 1 to a value outside of the stated range, the patient will still be eligible, and the weight should be rounded to the nearest value within the above range for dosing purposes.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 151 (Actual)
Dates: Start 2005-05; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (11):
- Spain (11):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Badajoz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Donostia / San Sebastian
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Espluges de Llobregat
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palma de Mallorca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sabadell
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sant Joan d'Alacant
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Cruz de Tenerife
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Terrassa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valencia

REFERENCES:
- [Derived] Bangs ME, Wietecha LA, Wang S, Buchanan AS, Kelsey DK. Meta-analysis of suicide-related behavior or ideation in child, adolescent, and adult patients treated with atomoxetine. J Child Adolesc Psychopharmacol. 2014 Oct;24(8):426-34. doi: 10.1089/cap.2014.0005. Epub 2014 Jul 14. PMID 25019647
- [Derived] Montoya A, Hervas A, Cardo E, Artigas J, Mardomingo MJ, Alda JA, Gastaminza X, Garcia-Polavieja MJ, Gilaberte I, Escobar R. Evaluation of atomoxetine for first-line treatment of newly diagnosed, treatment-naive children and adolescents with attention deficit/hyperactivity disorder. Curr Med Res Opin. 2009 Nov;25(11):2745-54. doi: 10.1185/03007990903316152. PMID 19785510
- [Derived] Escobar R, Montoya A, Polavieja P, Cardo E, Artigas J, Hervas A, Fuentes J. Evaluation of patients' and parents' quality of life in a randomized placebo-controlled atomoxetine study in attention-deficit/hyperactivity disorder. J Child Adolesc Psychopharmacol. 2009 Jun;19(3):253-63. doi: 10.1089/cap.2008.0109. PMID 19519260
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 158 patients enrolled during the Screening Period (Visits 1 and 2), but 7 did not receive study drug and are not included in the 151 patients randomized in the Double-Blind Period.
Groups:
- Atomoxetine: Double-Blind Acute Period: 0.5 mg/kg/day every day, by mouth for 2 weeks, 1.2 - 1.4 mg/kg/day every day, by mouth for 10 weeks Open-label Period: 1.2 - 1.4 mg/kg/day every day, by mouth for up to 1 year
- Placebo: Double-Blind Acute Period: every day, by mouth for 12 weeks,then possibility to switch to atomoxetine at 0.5 mg/kg/day every day, by mouth for 1 week Open-Label Period: 1.2 - 1.4 mg/kg/day every day, by mouth for up to 1 year
Period: Double-Blind Acute Treatment
Arm/Group | Atomoxetine | Placebo
Started | 100 | 51
Completed | 94 | 48
Not Completed | 6 | 3
Not completed — Parent's Decision | 3 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Non Protocol Compliance | 3 | 0
Not completed — Physician Decision | 0 | 2
Period: Open-Label Treatment Extension
Arm/Group | Atomoxetine | Placebo
Started | 94 | 48
Completed | 94 | 48
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atomoxetine | Placebo | Total
Number analyzed (Participants) | 100 | 51 | 151
Age Continuous [Mean (Standard Deviation); unit: years] | 10.3 (2.48) | 10.3 (2.43) | 10.3 (2.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 10 | 31
  Male | 79 | 41 | 120
Region of Enrollment [Number; unit: participants]
  Spain | 100 | 51 | 151
Attention-Deficit/Hyperactivity Disorder Subtype [Number; unit: participants]
  Inattentive | 30 | 19 | 49.0
  Hyperactive | 5 | 1 | 6.0
  Combined (Hyperactive-Inattentive) | 64 | 30 | 94.0
  Not Assessed | 1 | 1 | 2.0
Race/Ethnicity [Number; unit: participants]
  Caucasian | 98 | 47 | 145
  African | 0 | 1 | 1
  Hispanic | 2 | 3 | 5
Attention-Deficit/Hyperactivity Disorder Rating Scale-IV-Parent Version:Investigator-Administered [Mean (Standard Deviation); unit: units on a scale] — Measures the 18 symptoms contained in the Diagnostic and Statistical Manual of Mental Disorders Fourth Edition, Text Revision (DSM-IV-TR) diagnosis of Attention-Deficit/Hyperactivity Disorder. Individual item scores range from 0 (none/never or rarely) to 3 (severe/very often). Total scores range from 0 to 54.
  units on a scale | 39.1 (9.0) | 39.5 (9.0) | 39.2 (9.0)
Blood Pressure [Mean (Standard Deviation); unit: mmHg]
  Systolic Blood Pressure | 101.2 (10.01) | 100.5 (10.01) | 101.0 (9.98)
  Diastolic Blood Pressure | 57.9 (7.15) | 58.0 (7.68) | 57.9 (7.31)
Body Weight [Mean (Standard Deviation); unit: kilograms] | 37.9 (11.86) | 37.4 (12.18) | 37.7 (11.93)

OUTCOME MEASURES:

1. Primary Outcome: Attention-Deficit/Hyperactivity Disorder Rating Scale-IV-Parent Version:Investigator Administered and Scored (ADHDRS-IV-Parent:Inv) Total Score at 12 Week Endpoint
Description: Measures the 18 symptoms contained in the DSM-IV diagnosis of Attention-Deficit/Hyperactivity Disorder. Individual item scores range from 0 (none/never or rarely) to 3 (severe/very often). Total Scores range from 0 to 54.
Time Frame: Week 12
Population: Intention to Treat analysis. Single item missing scores were imputed with the mean score of the remaining items when computing subscale and total scores.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 99 | 50
units on a scale | 26.3 (12.7) | 34.8 (12.3)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mixed Model Repeated Measures analysis method: treatment, study site, visit, treatment-by-visit interaction, baseline, baseline-by-visit interaction; Mean Difference (Net) = -7.9, 95% CI [-11.0 to -4.8], Standard Error of Mean 1.6 — Least Squares Mean difference at week 12 (Atomoxetine minus Placebo)

2. Secondary Outcome: Attention-Deficit/Hyperactivity Disorder Rating Scale-IV-Parent Version:Investigator Administered and Scored (ADHDRS-IV-Parent:Inv) Total Score at 9 Weeks
Description: as for outcome 1
Time Frame: Week 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 99 | 50
units on a scale | 27.3 (12.3) | 34.4 (12.0)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; A gatekeeper strategy was employed for sequentially testing the secondary hypotheses using a REML-based Mixed-Model Repeated Measures (MMRM) technique as defined for the primary efficacy analyses. If primary hypothesis is significant at 0.05 (2-sided), first secondary hypothesis will be tested at Visit 6 from MMRM. If comparison is significant, subsequent secondary hypotheses will be tested in sequence until first null hypothesis fails to be rejected; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -6.5, 95% CI [-9.5 to -3.6], Standard Error of Mean 1.5 — Least Squares Mean difference at Week 9 (Atomoxetine - Placebo)

3. Secondary Outcome: Attention-Deficit/Hyperactivity Disorder Rating Scale-IV-Parent Version:Investigator Administered and Scored (ADHDRS-IV-Parent:Inv) Total Score at 6 Weeks
Description: as for outcome 1
Time Frame: Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 99 | 50
units on a scale | 28.7 (12.9) | 34.4 (12.0)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0009, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -5.2, 95% CI [-8.2 to -2.2], Standard Error of Mean 1.5 — Least Squares Mean difference at 6 weeks (Atomoxetine - Placebo)

4. Secondary Outcome: Attention-Deficit/Hyperactivity Disorder Rating Scale-IV-Parent Version:Investigator Administered and Scored (ADHDRS-IV-Parent:Inv) Total Score at 4 Weeks
Description: as for outcome 1
Time Frame: Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 99 | 50
units on a scale | 31.2 (12.0) | 35.5 (12.0)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0033, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -3.8, 95% CI [-6.4 to -1.3], Standard Error of Mean 1.3 — Least Squares Mean difference at 4 weeks (Atomoxetine - Placebo)

5. Secondary Outcome: Attention-Deficit/Hyperactivity Disorder Rating Scale-IV-Parent Version:Investigator Administered and Scored (ADHDRS-IV-Parent:Inv) Total Score Change From Week 6 to Week 12
Description: as for outcome 1
Time Frame: week 6 and week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 99 | 50
units on a scale
  Week 6 | 28.7 (12.9) | 34.4 (12.0)
  Week 12 | 26.3 (12.7) | 34.8 (12.3)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.013, Mixed Models Analysis — P-value is for the difference between groups in the change from 12 weeks minus 6 weeks; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -2.7, 95% CI [-4.9 to -0.6], Standard Error of Mean 1.1 — Least Squares Mean difference between groups (Atomoxetine - Placebo) in change from 6 weeks to 12 weeks

6. Secondary Outcome: Clinical Global Impressions- Attention-Deficit/Hyperactivity Disorder-Severity Changes From Baseline to Visit 7 (12 Weeks)
Description: Measures severity of the patient's overall severity of ADHD symptoms (1=normal, not at all ill; 7=among the most extremely ill patients).
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 99 | 50
units on a scale
  Baseline | 5.06 (0.93) | 5.04 (0.83)
  Week 12 | 3.89 (1.15) | 4.5 (0.91)

7. Secondary Outcome: Clinical Global Impressions- Attention-Deficit/Hyperactivity Disorder-Severity Change From Baseline to Endpoint (Visit 18) of the Open-Label Extension (107 Weeks)
Description: as for outcome 6
Time Frame: Baseline and Open-Label Endpoint (107 weeks)
Population: Intention to Treat analysis. Last observation carried forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Atomoxetine: 0.5 mg/kg/day QD, PO for 2 weeks, 1.2 - 1.4 mg/kg/day QD, PO for 10 weeks, then 1.2 - 1.4 mg/kg/day QD, PO for up to 1 year
Arm/Group | Atomoxetine
Number analyzed (Participants) | 140
units on a scale
  Baseline | 5.1 (0.92)
  Week 107 | 3.2 (1.28)

8. Secondary Outcome: Conners' Parent Rating Scale-Revised: Short Form (CPRS-R:S) Total Score Changes From Baseline to Endpoint (Week 12)
Description: The CPRS-R:S has 27 items to be completed by the parent to assess behavioral problems related to ADHD. Individual item scores range from 0 (not at all true/never/seldom: lowest impairment) to 3 (very much true/very often/very frequent: highest impairment). The total score is calculated as the sum of all items. Total scores range from 0 to 81.
Time Frame: Baseline and Week 12
Population: Intention to Treat analysis. Last observation carried forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 99 | 50
units on a scale
  Baseline | 54.6 (12.6) | 54.7 (13.6)
  Week 12 | 37.8 (18.7) | 48.5 (17.4)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value is for the difference between groups in the change from 12 weeks minus baseline; mixed model repeated measures analyis: treatment, visit, patient, and CPRS-R: S Total score at baseline as covariate, with treatment*visit interaction; Mean Difference (Net) = -10.7, 95% CI [-15.1 to -6.2], Standard Error of Mean 2.3 — Least Squares Mean difference between groups (Atomoxetine - Placebo) in change from baseline to 12 weeks

9. Secondary Outcome: Child Health and Illness Profile (CHIP) Change From Baseline to Endpoint (12 Weeks)
Description: Parent-rated assessment of a child's health status and level of functioning. It consists of 76 items. The majority of items assess frequency of activities or feelings using a five-point response format (for example, 'how good is your child at making friends?' 1=never, 5=always). Standard scores (t-value) were established, with all domains and subdomains having a mean score of 50 and standard deviation of 10. Standard scores are expressed in standard deviation units. T-score=[(Score-4.2382)*10/0.32835]+50. Higher scores mean improvement.
Time Frame: Baseline to 12 weeks
Population: Intention to Treat analysis. Last observation carried forward.
Measure: Mean (Standard Deviation); unit: standard deviation units
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 99 | 50
standard deviation units
  Parent: Satisfaction Baseline | 38.0 (14.9) | 39.0 (14.7)
  Parent: Comfort Baseline | 42.8 (12.5) | 44.4 (11.7)
  Parent: Resilience Baseline | 42.1 (11.2) | 41.8 (11.6)
  Parent: Risk Avoidance Baseline | 31.7 (15.8) | 34.1 (15.9)
  Parent: Achievement Baseline | 33.2 (9.5) | 33.1 (10.8)
  Parent: Satisfaction 12 Weeks | 40.4 (12.5) | 40.0 (13.8)
  Parent: Comfort 12 Weeks | 44.6 (11.4) | 44.1 (11.5)
  Parent: Resilience 12 Weeks | 45.3 (11.0) | 42.2 (10.8)
  Parent: Risk Avoidance 12 Weeks | 40.5 (14.8) | 35.9 (13.9)
  Parent: Achievement 12 Weeks | 38.0 (10.0) | 34.4 (10.3)
  Child/Adolescent: Satisfaction Baseline | 49.2 (9.2) | 50.0 (12.6)
  Child/Adolescent: Comfort Baseline | 49.9 (9.6) | 50.6 (7.9)
  Child/Adolescent: Resilience Baseline | 52.0 (10.8) | 52.0 (11.6)
  Child/Adolescent: Risk Avoidance Baseline | 47.6 (10.4) | 49.1 (11.3)
  Child/Adolescent: Achievement Baseline | 42.1 (10.3) | 44.6 (10.8)
  Child/Adolescent: Satisfaction 12 Weeks | 50.6 (9.2) | 52.3 (11.1)
  Child/Adolescent: Comfort 12 Weeks | 52.7 (8.2) | 51.9 (7.7)
  Child/Adolescent: Resilience 12 Weeks | 52.4 (9.5) | 52.2 (9.4)
  Child/Adolescent: Risk Avoidance 12 Weeks | 51.9 (8.7) | 49.7 (11.7)
  Child/Adolescent: Achievement 12 Weeks | 45.5 (10.2) | 45.7 (11.5)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; ANCOVA model: Dependent variable=standardized mean scores of domain at Visit 7 minus scores at Visit 1; Factors=Treatment, Investigator, Rater; Covariate=standardized mean scores of domain at Visit 1. Both treatment by rater and treatment by covariate interaction terms included in model; Test type: Superiority or Other; p = 0.810, ANCOVA — P-value for Parent: Satisfaction difference (Atomoxetine - Placebo) in the change from 12 weeks minus baseline; Mean Difference (Net) = 0.47, 95% CI [-3.39 to 4.33]
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.243, ANCOVA — P-value for Parent: Comfort difference (Atomoxetine - Placebo) in the change from 12 weeks minus baseline; Mean Difference (Net) = 1.96, 95% CI [-1.35 to 5.29]
Statistical Analysis 3: Comparison: Atomoxetine vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.419, ANCOVA — P-value for Parent: Resilience difference (Atomoxetine - Placebo) in the change from 12 weeks minus baseline; Mean Difference (Net) = 1.56, 95% CI [-2.26 to 5.39]
Statistical Analysis 4: Comparison: Atomoxetine vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for Parent:Risk Avoidance difference (Atomoxetine - Placebo) in the change from 12 weeks minus baseline; Mean Difference (Net) = 8.41, 95% CI [4.27 to 12.55]
Statistical Analysis 5: Comparison: Atomoxetine vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.042, ANCOVA — P-value for Parent:Achievement difference (Atomoxetine - Placebo) in the change from 12 weeks minus baseline; Mean Difference (Net) = 3.39, 95% CI [0.13 to 6.65]
Statistical Analysis 6: Comparison: Atomoxetine vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.323, ANCOVA — P-value for Child/Adolescent:Satisfaction difference (Atomoxetine - Placebo) in the change from 12 weeks minus baseline; Mean Difference (Net) = -1.36, 95% CI [-4.06 to 1.35]
Statistical Analysis 7: Comparison: Atomoxetine vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.452, ANCOVA — P-value for Child/Adolescent:Comfort difference (Atomoxetine - Placebo) in the change from 12 weeks minus baseline; Mean Difference (Net) = 0.92, 95% CI [-1.49 to 3.34]
Statistical Analysis 8: Comparison: Atomoxetine vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.910, ANCOVA — P-value for Child/Adolescent:Resilience difference (Atomoxetine - Placebo) in the change from 12 weeks minus baseline; Mean Difference (Net) = 0.16, 95% CI [-2.59 to 2.90]
Statistical Analysis 9: Comparison: Atomoxetine vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.006, ANCOVA — P-value for Child/Adolescent:Risk Avoidance difference (Atomoxetine - Placebo) in the change from 12 weeks minus baseline; Mean Difference (Net) = 3.56, 95% CI [1.04 to 6.08]
Statistical Analysis 10: Comparison: Atomoxetine vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.541, ANCOVA — P-value for Child/Adolescent:Achievement difference (Atomoxetine - Placebo) in the change from 12 weeks minus baseline; Mean Difference (Net) = 0.99, 95% CI [-2.21 to 4.19]

10. Secondary Outcome: Kiddie Schedule for Affective Disorders and Schizophrenia for School Aged Children-Present and Lifetime Version (K-SADS-PL)
Description: The K-SADS-PL is a semi-structured interview schedule for assessing psychiatric disorders in children and adolescents. It is used to assess the status of 32 DSM-IV child and adolescent psychiatric diagnosis.
Time Frame: Baseline
Population: Intention to Treat analysis. All randomized participants who took at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 99 | 50
participants
  Participants with any Comorbidity | 46 | 22
  Participants with Oppositional Defiant Disorder | 28 | 10
  Participants with Tic Disorder | 16 | 9
  Participants with Affective Disorders | 3 | 2
  Participants with Anxiety Disorders | 13 | 6
  Participants with Conduct Disorder | 0 | 0

11. Secondary Outcome: Attention-Deficit/Hyperactivity Disorder Rating Scale-IV-Parent Version:Investigator Administered and Scored (ADHDRS-IV-Parent:Inv) at 107 Weeks (Open-Label Extension)
Description: as for outcome 1
Time Frame: Week 107
Population: Intention to Treat analysis. Last observation carried forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 140
units on a scale | 21.4 (12.8)

12. Secondary Outcome: Vital Signs - Systolic Blood Pressure
Time Frame: Baseline and 12 weeks
Population: All randomized participants.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 100 | 51
mmHg
  Baseline | 98.7 (13.0) | 102.2 (11.4)
  12 Weeks | 102.9 (10.2) | 101.2 (11.7)

13. Secondary Outcome: Vital Signs - Diastolic Blood Pressure
Time Frame: Baseline and 12 weeks
Population: All randomized participants.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 100 | 51
mmHg
  Baseline | 56.4 (9.0) | 58.2 (7.2)
  12 Weeks | 59.3 (7.1) | 57.5 (8.6)

14. Secondary Outcome: Vital Signs - Pulse
Time Frame: Baseline and 12 weeks
Population: All randomized participants.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 100 | 51
beats per minute
  Baseline | 75.8 (9.8) | 77.0 (9.3)
  12 Weeks | 84.5 (12.5) | 79.0 (9.7)

15. Secondary Outcome: Vital Signs - Weight
Time Frame: Baseline and 12 weeks
Population: All randomized participants.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 100 | 51
kilograms
  Baseline | 38.0 (12.0) | 37.5 (12.3)
  12 Weeks | 37.0 (11.5) | 38.9 (12.8)

ADVERSE EVENTS:
Arm/Group | Atomoxetine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/100 | 1/51
Other Adverse Events (participants affected / at risk) | 80/100 | 38/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine (N=100) | Placebo (N=51)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine (N=100) | Placebo (N=51)
Tachycardia (Cardiac disorders) | 4 (4) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 17 (20) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 6 (7) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 3 (3)
Nausea (Gastrointestinal disorders) | 5 (7) | 2 (2)
Vomiting (Gastrointestinal disorders) | 14 (22) | 7 (7)
Fatigue (General disorders) | 10 (11) | 1 (1)
Pyrexia (General disorders) | 7 (8) | 3 (3)
Ear infection (Infections and infestations) | 0 (0) | 3 (3)
Nasopharyngitis (Infections and infestations) | 7 (8) | 5 (7)
Decreased appetite (Metabolism and nutrition disorders) | 31 (31) | 4 (4)
Dizziness (Nervous system disorders) | 7 (8) | 2 (2)
Headache (Nervous system disorders) | 24 (29) | 7 (8)
Somnolence (Nervous system disorders) | 23 (24) | 2 (2)
Irritability (Psychiatric disorders) | 14 (16) | 5 (6)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days